CLINICAL TRIAL: NCT02107326
Title: Webdia Study: Use of Smartphones to Improve Diabetes Control and Quality of Life in Children With Type 1 Diabetes
Brief Title: Randomized Crossover Study to Test the Impact of Using a Software for Smartphones and Tablets in Treating Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philippe Klee (Other)
Responsible Party: Sponsor-Investigator, Philippe Klee, MD-PhD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CER13-272
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Type 1 Diabetes; Quality of Life; Hypoglycaemia
Keywords: Type 1 diabetes; HbA1C; Quality of Life; Hypoglycaemia; Self-management; Telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Webdia Software use (Experimental): Use of Webdia Software during 3 months by the patient. Monthly review of blood glucose values by the medical team and automatic adjustment of insulin doses by the team.
  Interventions: Device: Webdia Software
- Observation (No Intervention): No use of the software. No intervention.

INTERVENTIONS:
Device: Webdia Software
  Arms: Webdia Software use

SUMMARY:
The purpose of this study is to evaluate the impact of a software for smartphones and tablets on type 1 diabetes control and quality of life

DETAILED DESCRIPTION:
The hypothesis underlying this project, is that most calculations necessary for flexible intensive insulin therapy for type 1 diabetes in children can be performed using software installed on a smartphone or tablet that nowadays is carried by most parents and children. Smartphones and tablets can easily communicate with each other and with a desktop computer via the Internet, thereby permitting the exchange of information such as blood glucose values or types of meals among family members and physicians. Finally, software collecting blood glucose values and merging values obtained on different devices easily permits reviewing these values by the patient and sending them to the physician's office, thereby avoiding consultations during which no blood glucose values are brought by the patient.

We hypothesize that the Webdia software, that will be tested in this randomized crossover study, will increase treatment compliance and therefore will improve diabetes self-management. We believe, the software will facilitate the adaptation of insulin schemes by physicians and therefore will lead to improved HbA1C values. We also think that this software will improve the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 - 18 years
* Type 1 diabetes mellitus with positive auto-antibodies against Islet Antigen (IA) 2, insulin, islets, Glutamic Acid Decarboxylase (GAD) 65 or Zink
* Disease duration equal or more than 6 months
* Treatment by subcutaneous insulin: by multiple daily injections of pump therapy

Exclusion Criteria:

* Previous use of Webdia Software
* Absence of hardware necessary to install the Webdia Software

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2014-05; Primary Completion 2017-08-15 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Effect of Webdia Software use on HbA1C | 0, 3, 6 and 9 months after inclusion

SECONDARY OUTCOMES:
Effect of Webdia Software use on quality of life | 0, 3, 6 and 9 months after inclusion
  Quality of life assessment by the use of the Diabetes Quality of Life for Youths (DQOLY) questionnaire published by Ingersoll et al. 1991.
Effect of Webdia Software use on the incidence of hypoglycaemic events | During 2 weeks at the end of the 3-months period of Webdia Software use

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Klee, MD-PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland